CLINICAL TRIAL: NCT06822686
Title: Assessment of the Feasibility of Autologous Bone Marrow-derived Mesenchymal Stem Cells in the Management of Fistulating Perianal Crohn's Disease
Brief Title: Autologous Stem Cells in the Management of Fistulating Perianal Crohn's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Mark Bignell, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Stemcell
Record Dates: First submitted 2023-12-20; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Fistula in Ano; Crohn Disease
Keywords: Stem cell
MeSH Terms: conditions — Rectal Fistula; Crohn Disease

STUDY DESIGN:
Intervention Model Description: Feasibility trial to assess the use of autologous stem cells in the management of fistulating perianal Crohn's. Observational study. No Comparator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Injection of stem cell into fistulating perianal Crohn's disease (Experimental): At surgery participants will undergo an examination of the anorectum under anaesthesia and if suitable the stem cells will be harvested. Harvest of the bone marrow-derived mesenchymal stem cells is performed by aspirating 60ml of bone marrow. The aspirate is then centrifuged in theatre and the mesenchymal stem cells prepared in theatre by a representative from (Synergy Medical Technologies). Once prepared they are administered immediately into and around the fistula tract. The internal opening is then closed.
  If the participant is not suitable they will undergo best surgical practice and will be excluded from the study. They will then undergo follow-up as dictated by their clinical condition.
  All participants will undergo the procedure as a day case.
  Interventions: Device: Harvest and injection of stem cells

INTERVENTIONS:
Device: Harvest and injection of stem cells — Stem cells will be harvested from bone marrow aspirate and injected into the fistula tract The stem cells are the device intervention for this trial and we are looking to assess the procedure of harvesting and injecting the stem cells Patients will undergo study questionnaire: Harvey-Bradshaw Index, perianal Crohn's disease activity index, and Short IBD questionnaire will be administered before surgery and then at 6 weeks, 3 and 6 months after stem cell intervention.

SUMMARY:
Crohn's disease is a chronic inflammatory condition that can affect any part of the bowel which can be controlled by a combination of medical and surgical treatments but cannot be cured. A 1/3 of patients have involvement of the perianal region. There are several conditions that can affect the perianal region but the most debilitating is the presence of fistulating disease. Fistulae are small tunnels that run under the skin from the inside of the anus to skin outside the anus and are associated with the inflammatory process seen with Crohn's disease. They can cause pain, infection and discharge which adversely affects the quality of life of the patient. Surgery can be used to treat the symptoms however cure is often difficult to achieve.

Stem cells have anti-inflammatory potential and have been shown to be a useful treatment for this condition in combination with effective medical therapy. The stem cells used in the studies need to be prepared 48 hours before use which limits their usage and this is not readily available in the UK.

The proposed study aims to assess the feasibility of using autologous stem cells prepared with a rapid preparation system at the time of surgery, within the operating room (currently in use at Oxford University Hospitals NHS Foundation Trust (OUH) within the orthopaedic department for a different indication) for fistulating anal Crohn's disease. The stem cells are derived from the patients own bone marrow. The patients undergoing surgery would be having it done for the stem cell treatment. They will then undergo 3 follow up visits and complete questionnaires at each visit alongside a clinical assessment. This study is funded by Occtopus (Colorectal charity based in Oxford).

DETAILED DESCRIPTION:
This is a singe-centre interventional study to assess the feasibility of administering autologous bone marrow-derived mesenchymal stem cells to promote healing of fistulating perianal Crohn's disease after medical optimisation (i.e their luminal disease is well controlled by medical therapy which is at its optimum dosing as determined by the gastroenterology team). It will be conducted in tertiary care by surgeons who are experienced in managing this condition. Participants will be identified and their suitability assessed for entry into the study. Participants will have had a MRI Rectum prior to inclusion as this is a standard radiological modality to assess and managing this condition in clinical practice. Participants may have undergone an examination of their anorectum under anaesthesia in their initial work-up however this is not necessary for inclusion into the trial. If eligibility criteria are met and the patient wishes to proceed then a follow-up appointment will be made to consent them into the study. Participants will undergo surgery and at this stage the stem cells will be harvested and then injected into the fistula tract. Participants will be assessed at regular intervals post-intervention.

The study involves 2 screening visits, 1 intervention visit (surgery) and 3 post-intervention visits; a total of 6 visits. The study does involve an increase in clinic appointments compared to routine post-operative care. These participants are normally seen routinely in clinic with a frequency of 6 weeks to 6 monthly depending on the severity of the symptoms. It would be anticipated the participants enrolled into the trial would usually be seen 2-4 times over the same period if they were not involved in the trial.

At the visits a clinical record form will be completed by the surgeon in charge of their care which records baseline demographic data as well as clinical assessment of the fistula. Data will be entered in this record at each visit. Questionnaires assessing disease activity (Harvey-Bradshaw Index (HBI) and Perianal Crohn's Disease Activity Index (PCDAI)) and QoL (Short IBD) are administered at the second screening visit and at the 6 week and 3 months visits (PCDAI) and at 6 months (HBI, PCDAI, and SIBD). The outpatient nurses will administer the questionnaires and these will be completed before the participant sees the surgeon. This is a normal process within the outpatient department and will not require any training for the outpatient nurses. The questionnaires will be collected by the surgeon who will ensure they are complete. At the operation details of the operation will be recorded on the Clinical Record File (as well as an operation note on the electronic patient record held by OUH NHS Trust). The WHO checklist will also be completed. This is a mandatory requirement for all theatre cases. The checklist allows for a debrief at the end of each case and information regarding the procedure will be included here. A copy of this will be incorporated into the clinical record file.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with perianal Crohn's disease
* Medically controlled proximal disease as confirmed by endoscopy or Harvey Bradshaw Index scores of less than 7 (remission / mild disease)
* Recent MRI scan to assess fistulating perianal Crohn's
* Non-branching fistula with no more than 1 internal opening and 2 external opening i.e. a single tract.
* No previous definitive fistula treatment (seton excluded)
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.
* Ongoing perianal sepsis or anal stenosis
* Patients with a defunctioning stoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using autologous mesenchymal stem cells in the management of fistulating perianal Crohn's disease. | During surgery
  Operative time and difficulties encountered intraoperatively will be documented on the operation note. Subjective impression of the operating surgeon alongside feedback from the nursing team in theatre will help assess the procedure. Feedback from the operative team will be documented on the WHO checklist (where a section for feedback exists).

SECONDARY OUTCOMES:
Safety of stem cell treatment | after surgery for 6 months with clinical review at 6 weeks, 3 months and 6 months
  patient reported adverse effects and clinical assessment
Safety of stem cell treatment | after surgery for 6 months with clinical review at 6 weeks, 3 months and 6 months
  Changes in Quality of life or Disease activity scores (monitored by perianal Crohn's disease activity index, Harvey-Bradshaw Index, and Short IBD questionnaires)
Safety of stem cell treatment | after surgery for 6 months with clinical review at 6 weeks, 3 months and 6 months
  Attendance to Emergency department
Safety of stem cell treatment | after surgery for 6 months with clinical review at 6 weeks, 3 months and 6 months
  Contact with IBD nurse specialists

IPD SHARING:
Plan to Share IPD: No